CLINICAL TRIAL: NCT04618250
Title: A Cluster Randomized, Pilot Trial of Coordinated, Co-produced Care to Reduce Excess Mortality and Improve Quality of Life in Patients With Severe Mental Illness in General Practice Setting
Brief Title: Improving Physical Health in Patients With Psychiatric Disorders in General Practice (SOFIA)
Acronym: SOFIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Susanne Reventlow, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NNF16OC0022038
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Psychiatric Disorder; Schizophrenia; Bipolar Disorder; Severe Depression
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coordinated, co-produced health care (Experimental)
  Interventions: Other: SOFIA model
- Care as usual (No Intervention): Care as usual

INTERVENTIONS:
Other: SOFIA model — A mandatory two day course for general practitioners assigned to the intervention group A prolonged consultation at the general practitioner Use of an individual care plan
  Arms: Coordinated, co-produced health care

SUMMARY:
People with a severe mental illness (SMI) have an increased risk for premature mortality, predominantly due somatic health conditions. Evidence indicates that prevention and improved treatment of somatic conditions in patients with SMI could reduce this excess mortality. This paper reports a protocol designed to evaluate the feasibility and acceptability of a coordinated co-produced care programme (SOFIA model) in the general practice setting to reduce mortality and improve quality of life in patients with severe mental illness. The primary outcomes are description of study feasibility (recruitment and retention) and acceptability.

The SOFIA trial is designed as cluster randomized controlled trial targeting general practices in two regions in Denmark. 12 practices will each recruit 15 community-dwelling patients aged 18 and older with severe mental illness (SMI). Practices will be randomized in a ratio 2:1 to deliver a coordinated care program or care-as-usual during a 6 month period. An online randomized algorithm is used to perform randomization. The coordinated care program comprises enhanced educational training of general practitioners and their clinical staff, and prolonged consultations focusing on individual needs and preferences of the patient with SMI. Assessments are administered at baseline, and at end of study period.

If delivery of the intervention in the general practice setting proves feasible, a future definitive trial to determine the effectiveness of the intervention in reducing mortality and improving quality of life in patients with SMI can take place.

ELIGIBILITY:
Inclusion Criteria:

* Registered at a general practice situated in the Danish Capital Region or the Region of Zealand;
* Registered at general practice with International Classification of Primary Care version 2 (ICPC-2) diagnostic code p72 (psychotic disorders);
* Registered at general practice with ICPC-2 diagnostic code p73 (bipolar mood disorders);
* Prescription of Lithium (Anatomical Therapeutic Chemical (ATC): N05AN);
* Registered at general practice with ICPC-2 diagnostic code p76 AND (Prescription of Lamotrigine (N03A09) OR Carbamazepine (N03AF01) OR Valproic Acid (N03AG01));
* Registered at general practice with ICPC-2 diagnostic code p76 (unipolar depressive disorders) AND (Prescription of tricyclic antidepressants (N06AA) AND/OR venlafaxine (N06AX16) AND/OR duloxetine (N06AX21) AND/OR Monoamine Oxidase A Inhibitor (MAOi) (N06AG) AND/OR non-selective MAOi (N06AF)).

Exclusion Criteria:

* Subjected to any type of legal measure as stipulated in the Danish Mental Health Law;
* Registered with a dementia diagnosis ICPC-2 p70 (dementia);
* Receiving end-of-life care;
* Non-Danish speakers;
* Assumed by the patient's general practitioner to have an overall functional level that is too low for meaningful participation in trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the design in terms of recruitment of practices and patients | 6 months after randomization
  Proportion of contacted general practices, which agree to participate in the study and the eligibility and consent rate of patients.
Acceptability of the intervention for patients and general practitioners, staff and patients. | Entire study period (6 months)
  Qualitative semi-structured interviews with patients and general practitioners, staff and patients.
Retention of patients during the study | 6 months after randomization
  Proportion of recruited patients in the intervention group who attend the first consultation.
Acceptability of REDcap software for general practitioners | Entire study period (6 months)
  Qualitative semi-structured interviews with general practitioners.
Effectiveness of the collecting Multimorbidity Questionnaires | 6 months after randomization
  Proportion of returned and completed Multimorbidity Questionnaires.
Effectiveness of the collecting EQ5D-5L questionnaires | 6 months after randomization
  Proportion of returned and completed EQ5D-5L questionnaire.
Mortality | 6 months after randomization
  Number of all-cause deaths of participants during the 6 month trial period.
Hospitalizations | 6 months after randomization
  Number of all-cause in- and outpatient hospitalizations of participants during the 6 months trial period.

SECONDARY OUTCOMES:
Multimorbidity Questionnaires (MMQ) scores | 3 times during study period (at baseline, before prolonged consultation and 6 months after randomization
  Scores on Multimorbidity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Reventlow, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Participants' study information will not be released outside of the study without the written permission of the participant.

REFERENCES:
- [Derived] Tranberg K, Due TD, Rozing M, Jonsson ABR, Kousgaard MB, Moller A. Challenges in reaching patients with severe mental illness for trials in general practice-a convergent mixed methods study based on the SOFIA pilot trial. Pilot Feasibility Stud. 2023 Oct 31;9(1):182. doi: 10.1186/s40814-023-01395-y. PMID 37908003
- [Derived] Tranberg K, Jonsson A, Due T, Siersma V, Brodersen JB, Bissenbakker K, Martiny F, Davidsen A, Kjellberg PK, Doherty K, Mercer SW, Nielsen MH, Reventlow S, Moller A, Rozing M; SOFIA Study Group. The SOFIA pilot study: assessing feasibility and fidelity of coordinated care to reduce excess mortality and increase quality of life in patients with severe mental illness in a general practice setting; a cluster-randomised pilot trial. BMC Prim Care. 2023 Sep 16;24(1):188. doi: 10.1186/s12875-023-02141-2. PMID 37715123
- [Derived] Rozing MP, Jonsson A, Koster-Rasmussen R, Due TD, Brodersen J, Bissenbakker KH, Siersma V, Mercer SW, Guassora AD, Kjellberg J, Kjellberg PK, Nielsen MH, Christensen I, Bardram JE, Martiny F, Moller A, Reventlow S; SOFIA Study Group. The SOFIA pilot trial: a cluster-randomized trial of coordinated, co-produced care to reduce mortality and improve quality of life in people with severe mental illness in the general practice setting. Pilot Feasibility Stud. 2021 Sep 3;7(1):168. doi: 10.1186/s40814-021-00906-z. PMID 34479646